CLINICAL TRIAL: NCT04866498
Title: Pharmacotherapy Personalization of Cancer Patients Based on Modern Analytical and Computational Techniques
Brief Title: Pharmacotherapy Personalization of Cancer Patients
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: The Greater Poland Cancer Centre (Other); Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Agnieszka Bienert, Full Professor, Poznan University of Medical Sciences
Other Study IDs: 763/2016; 2015/17/B/NZ7/03032 (Other Grant/Funding Number: Polish National Science Centre)
Record Dates: First submitted 2021-04-21; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Head and Neck Neoplasms; Oncologic Patients
Keywords: Anesthesia; Intensive Care Units; Pharmacokinetics; Pharmacodynamics; Surgical patients; Analgosedation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Infusions, Intravenous; Analgesics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Analgosedation in ICU patients after head and neck tumor resection in general anesthesia: Head and neck tumor resections were performed in general anesthesia. Midazolam and etomidate or propofol were used in introduction and then anesthesia was maintenance with sevoflurane. Patients received intravenous continuous infusion of oxycodone as an analgesic component and sedatives (propofol/dexmedetomidine/midazolam) during analgosedation in ICU.
  Interventions: Drug: Infusion Intravenous

INTERVENTIONS:
Drug: Infusion Intravenous
  Other Names: Analgesics and sedatives intravenous continuous infusion

SUMMARY:
Treatment personalization could ensure better outcome than standard procedures. It is particularly important in intensive care units where patients received many drugs and procedures. Their health status can change very fast. The oncologic patients treated in intensive care units are a special group of patients. Factors related to cancer influence extra their health status. The aim of this study is population pharmacokinetic-pharmacodynamic analysis drugs that are routinely used during an analgosedation in ICU oncologic patients. Analgosedation is monitored by drugs plasma concentration, the depth of sedation (bispectral index) and vital parameters like: systolic and diastolic blood pressure, mean arterial pressure, heart rate. Moreover, the TNM Staging System, biochemical parameters, The American Society of Anesthesiologists (ASA) physical status classification will be checked like potential factors influencing on pharmacokinetics and pharmacodynamics drugs used in the study.

DETAILED DESCRIPTION:
The oncologic patients are qualified to head and neck tumor resection in general anesthesia. The anesthesia introduction is performed with single dose of midazolam, fentanyl, rocuronium and propofol/etomidate. Sevoflurane is used in anesthesia maintenance. Patients are transported to ICU after operation. Then they are kept for several hours in analgosedation. All used drugs are given by intravenous continuous infusion. Oxycodone is an analgesic component of analgosedation. Midazolam, dexmedetomidine and/or propofol are used as sedatives (2-3 drugs in every patient). Whole blood samples (2.0 ml) are collected during the study to measure drugs concentrations - 3-4 times during infusion, 5, 10, 15, 30, 60 minutes and 2, 4, 6 hours after the infusion cessation. Vital parameters and bispectral index are monitored during analgosedation and 6 hours after the infusion cessation and noted every 15-60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old,
* qualifications to oncologic surgery,
* needing of analgosedation in ICU after an operation

Exclusion Criteria:

* proven allergies to used in anesthetics or/analgosedation medicaments,
* lack of written confirmed consent of a patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The adult patients with recognition of head and neck tumor who are qualified to tumor resection in general anesthesia and needing analgosedation in ICU after operation.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Measurement of the depth of sedation using bispectral index | from the beginning of analgosedation to 6 hours after analgosedation
  Continuous measurement of the depth of sedation using bispectral index during analgosedation in intensive care unit.

SECONDARY OUTCOMES:
Oxycodone plasma concentrations [ng/ml] | 3-4 times during infusion, 5, 10, 15, 30, 60 minutes and 2, 4, 6 hours after the infusion cessation
  Measurements of oxycodone and noroxycodone plasma concentrations [ng/ml] during and after analgosedation. Whole blood samples (2.0 ml) were collected according to the study protocol.
Dexmedetomidine plasma concentrations [ng/ml] | 3-4 times during infusion, 5, 10, 15, 30, 60 minutes and 2, 4, 6 hours after the infusion cessation
  Measurements of dexmedetomidine plasma concentrations [ng/ml] during and after analgosedation. Whole blood samples (2.0 ml) were collected according to the study protocol.
Midazolam plasma concentrations [ng/ml] | 3-4 times during infusion, 5, 10, 15, 30, 60 minutes and 2, 4, 6 hours after the infusion cessation
  Measurements of midazolam and alfa-hydroxymidazolam plasma concentrations [ng/ml] during and after analgosedation. Whole blood samples (2.0 ml) were collected according to the study protocol.
Propofol plasma concentrations [ng/ml] | 3-4 times during infusion, 5, 10, 15, 30, 60 minutes and 2, 4, 6 hours after the infusion cessation
  Measurements of propofol plasma concentrations [ng/ml] during and after analgosedation. Whole blood samples (2.0 ml) were collected according to the study protocol.
Systolic blood pressure | before the beginning of analgosedation, during analgosedation, up to 6 hours after analgosedation
  Measurements of systolic blood pressure during analgosedation in intensive care unit.
Diastolic blood pressure | before the beginning of analgosedation, during analgosedation, up to 6 hours after analgosedation
  Measurements of diastolic blood pressure during analgosedation in intensive care unit.
Heart rate | before the beginning of analgosedation, during analgosedation, up to 6 hours after analgosedation
  Measurements of heart rate during analgosedation in intensive care unit.
Mean arterial pressure | before the beginning of analgosedation, during analgosedation, up to 6 hours after analgosedation
  Measurements of mean arterial pressure during analgosedation in intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Bienert, MSC, PhD, Principal Investigator — Poznan University of Medical Sciences; Edmund Grzeskowiak, MSC, PhD, Study Director — Poznan University of Medical Sciences
Locations (2):
- Poland (2):
  - Greater Poland Cancer Centre, Poznan, Greater Poland Voivodeship
  - Medical University of Gdansk, Gdansk, Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
pharmacokinetic and pharmacodynamic data (concentration/effect/time profiles) of individuals will be available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available in 6-12 months and available for 5 years
Access Criteria: Scientists